CLINICAL TRIAL: NCT01014858
Title: Multi-centre UK Study of the Acetylcholinesterase Inhibitor Donepezil in Early Dementia Associated With Parkinson's Disease
Acronym: MUSTARDD-PD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to low recruitment
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: University of Newcastle Upon-Tyne (Other); University of Cambridge (Other); University of Manchester (Other); University of Birmingham (Other); Bangor University (Other); London School of Economics and Political Science (Other); University College, London (Other); Lancashire Care NHS Foundation Trust (Network); Newcastle University (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5137; 08/13/14 (Other Grant/Funding Number: NIHR Health Technology Assessment Programme 08/13/14)
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; mild dementia; donepezil; NIHR HTA
MeSH Terms: conditions — Parkinson Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donepezil (Experimental): 5mg of Donepezil for the first 8 weeks raising to 10mg thereafter if patient adjusted to 5mg dose. 10mg does continues for the remainder of the study.
  Interventions: Drug: Donepezil
- Placebo (Placebo Comparator): Patient commences medication to match appearance of 5mg donepezil for first 8 weeks then 10mg for the remainder of the study.
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — 5mg donepezil daily for first 8 weeks and then increased to 10mg daily for the remainder of the study.

SUMMARY:
To demonstrate the superiority of donepezil over placebo in improving cognitive function, neuropsychiatric burden and functional ability in people with Parkinson's disease and mild dementia after 24 months of treatment.

To demonstrate the superiority of donepezil over placebo in improving patient and carer quality of life and to establish the cost-effectiveness of donepezil.

To determine the instrument most suitable for evaluating change in cognition in people with Parkinson's disease and mild dementia.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of Parkinson's disease according to UK Parkinson's Disease Society Brain Bank Criteria. These criteria are in standard use throughout the NHS in the UK and were supported by the NICE guidelines.
2. People with mild dementia associated with PD, where the patient and/or their family have become aware of cognitive with or without behavioural symptoms that are causing functional impairment. "Dementia" will be defined according to recently published Movement Disorder Society Task Force criteria for dementia associated with Parkinson's Disease and "operationalised" using the Addenbrooke's Cognitive Examination (ACE-R). The ACE-R permits some description of the dementia profile and also quantifies global impairment. It is increasingly used by clinicians in the UK to identify demented subjects, is relatively quick to perform (15 minutes or so), requires no specific training and produces a total score (0-100), from which the MMSE (0-30) can also be extracted. Participants will have an ACE-R of 88 or less. If this criterion is met, subjects will be further assessed using the Mattis Dementia Rating Scale (DRS-2). An age- and education-corrected total DRS-2 score of less than 8 but greater than 4 (corresponding to between the 6th and 28th percentile) will be used to define "mild" dementia".
3. Community-living and a spouse, close relative or well established carer to accompany the subject to act as an informant.
4. Where relevant, women of child bearing potential must be using adequate contraception for duration of study.

Exclusion Criteria:

1. Dementia that develops within one year of the onset of motor symptoms. The reason for this "one year rule" is to specifically exclude participants with Dementia with Lewy Bodies (DLB). This exclusion criterion is consistent with recommendations made in the Movement Disorder Society Dementia Task Force Diagnostic Criteria and the Third Report of the DLB Consortium.
2. People with such severe motor disability, or who are so impaired in their activities of daily living from other aspects of their PD, that it would interfere with cognitive and global assessments.
3. Severe current depressive episode. Low mood may impact upon accurate cognitive assessment and major depression is therefore listed as a feature which, when present, makes it impossible to reliably diagnose PDD in the Movement disorder Society Task Force PDD Criteria. This will be operationalised using the self-completed Beck Depression Inventory and a cut-off score of 13, as recommended by a recent Movement Disorder Society Task Force report. The BDI score is considered robust in the face of mild to moderate cognitive impairment.
4. Unstable significant medical co-morbidity.
5. Patient receiving an anticholinergic drug for control of parkinsonian motor symptoms.
6. Previous exposure to a cholinesterase inhibitor
7. Presence of a condition that is contraindicative to use of donepezil (including a clinically significant cardiac conduction defect found in patient history or from screening ECG); see SmPC (Appendix W) for details.
8. Allergy/hypersensitivity to excipients of donepezil or placebo
9. Patient receiving the N-methyl-d-aspartate antagonist memantine.
10. Previous neurosurgery for Parkinson's disease. This will apply to only a small minority of predominantly younger cases. The main reason for this exclusion relates to ongoing uncertainty over the potential confounding effects of deep brain stimulation upon both mood and cognition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate the superiority of donepezil over placebo in improving cognitive function, neuropsychiatric burden and functional ability in people with Parkinson's disease and mild dementia after 24 months of treatment. | After 24 month of treatment

SECONDARY OUTCOMES:
To demonstrate the superiority of donepezil over placebo in improving patient and carer quality of life and to establish the cost-effectiveness of donepezil. | 26, 52 and 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David J Burn, Professor, Study Chair — Newcastle University; Roger A Barker, Dr, Study Director — Cambridge University; Belinda Braithwaite, Mrs, Study Director — lay person; Alistair Burns, Professor, Study Director — School of Community Based Medicine, University of Manchester; Carl E Clarke, Professor, Study Director — Clarke; Elaine McColl, Professor, Study Director — University of Newcastle Upon-Tyne; John V Hindle, Dr, Study Director — Llandudno Hospital & University of College Wales; Martin Knapp, Professor, Study Director — London School of Economics and Political Science; Andrew J Lees, Professor, Study Director — University College, London; Iracema Leroi, DR, Study Director — Lancashire Care Trust, Royal Blackburn Hospital; Ian G McKeith, Professor, Study Director — Newcastle University; John T O'Brien, Professor, Study Director — Newcastle University; Keith Wheatley, Professor, Study Director — Cancer Research UK Clinical Trials Unit, School of Cancer Sciences, University of Birmingham; Ian N Steen, Dr, Study Director — University of Newcastle Upon-Tyne; Jennifer Wilkinson, Mrs, Study Director — University of Newcastle Upon-Tyne; Sharon Erb, Mrs, Study Director — University of Newcastle Upon-Tyne; Daniel Weintraub, Study Director — Associate Professor of Psychiatry and Neurology, Perelman School of Medicine at the University of Pennsylvania; Lynn Rochester, Study Director — Professor of Human Movement Science, Institute for Ageing and Health, Newcastle University
Locations (22):
- United Kingdom (22):
  - Newcastle, Newcastle upon Tyne, Tyne and Wear
  - Royal United Hospital (RUH) Bath NHS, Bath
  - Sandwell and West Birmingham NHS Foundation Trust, Birmingham
  - Steps and Pines, Southmead Hospital, Bristol
  - Pennine Acute Hospitals NHS Trust, Bury
  - Cambridge Centre for Brain Repair, Cambridge
  - Dr Lakmali Sugathapala, Derby
  - Royal Bournemouth & Christchurch Hospitals NHS Foundation Trust, Dorset
  - NHS Greater Glasgow and Clyde, Glasgow
  - Dr Pippa Metcalf, Gloucester
  - Llandudno Hospital, Betsi Cadwaladr University Health Board & School of Medical Sciences, Llandudno
  - King's College Hospital NHS Foundtion Trust, London
  - Manchester Mental Health & Social Care NHS Trust, Manchester
  - Milton Keynes, Milton Keynes
  - Royal Gwent Hospital, Newport
  - North Tyneside General Hospital, Northumberland
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Plymouth Hospitals NHS Trust, Plymouth
  - Poole Hospital NHS Trust, Poole
  - Southampton General Hospital, Southampton
  - Dr Dhakam, Surrey